CLINICAL TRIAL: NCT04256720
Title: The Clustering of Lifestyle Behaviours in a Multi-ethnic Population: A Questionnaire Study
Brief Title: The Multi-Ethnic Lifestyle Study
Acronym: MELS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0672
Record Dates: First submitted 2018-10-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus; Chronic Kidney Diseases; Cardiovascular Diseases; Obstructive Sleep Apnea; Respiratory Disease; Cancer; Stroke; Chronic Pain; Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse); Healthy
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Cardiovascular Diseases; Sleep Apnea, Obstructive; Respiration Disorders; Neoplasms; Stroke; Chronic Pain; Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: No intervention — No intervention - questionnaire study

SUMMARY:
The study design is cross-sectional using a self-completion questionnaire in an English speaking multi-ethic population within Leicester and Leicestershire. The study will adopt a convenient and purposive sampling recruitment strategy across a variety of settings within Leicestershire to facilitate recruitment of a wide range of participants.

DETAILED DESCRIPTION:
It is well reported that lifestyle behaviours can play a significant role in health, contributing towards chronic disease and mortality. The World Health Organisation (WHO) describes behavioural risk factors as 'the epidemic of the 21st Century', defining a strategic objective to not only promote health and development, but to prevent and reduce health conditions associated with behavioural risk factors such as smoking, alcohol consumption, unhealthy diets and poor physical activity (1).

In England, reports by the Department of Health (DoH) have identified significant concerns in national attitudes towards health stating that 60% of the adult population hold a negative or fatalistic attitude towards their own health, and that these attitudes are particularly prominent in disadvantaged groups (2). This has been corroborated in recent statistics published this year by Public Health England (PHE) comparing the health status in local authorities with that of the wider population, reporting that in the total for England, 15.5% of the population are active smokers, 35.1% are not physically active (a figure likely to be much higher with the use of objective measures), and 64.8% demonstrate excessive body weight.

When comparing Leicester (reported as one of the 20% most deprived districts in the UK) with this national average, smoking and weight statistics are seen as on par with the wider population benchmark, with significantly lower levels of physical activity (50%), significantly higher rates of reported diabetes (8.9%), and significantly lower life expectancy in both men and women (77.1 and 81.6 years) (3). Leicester is an ethnically diverse city, with a high population of South Asians, who have been shown to be substantially less physically active compared to the national average (4-6), which may contribute to the statistics seen in the city's public health profile. When looking at the same health report for Leicestershire county, reported as one of the 20% least deprived counties in England, the statistics demonstrate that the health of people is proportionally better than that of the wider population average, with only recorded diabetes shown as below the England average, and all other factors reported as either the same or significantly better in comparison, highlighting the potential impact of socioeconomic disparity in health outcomes (7).

An important lifestyle behaviour that is can often be discounted when considering health statistics is sleep and chronotype. Insufficient sleep has been shown to have significant impacts on physical health with multiple large meta-analyses demonstrating associations with obesity and cardiometabolic disease (8-11). These findings have been corroborated by large UK surveys demonstrating that inadequate sleep is associated with increased BMI and poor metabolic profiles (12), as well as increased cardiovascular disease and type 2 diabetes (13). A longitudinal study in the UK also demonstrated links between insufficient sleep with psychological health problems including depression, anxiety and increased experiences of pain (14). An individual's chronotype, understood as a behavioural trait determined by their circadian rhythm to be either morning- or evening orientated, has shown a number of associated health implications. Research has shown that being a "night owl", as opposed to an "early bird", increases the likelihood of a number of physical and psychological health concerns including mood and anxiety disorders, personality disorders, substance misuse, insomnia, sleep apnoea, arterial hypertension, bronchial asthma, type 2 diabetes, and infertility, with an overall lower mortality (15).

While there has been extensive data on the impact of single lifestyle behaviours on disease related outcomes and mortality, the evidence on combined effects of lifestyle behaviours has not received the same attention, although the available data is compelling. In a systematic review and meta-analysis exploring lifestyle factors related to all-cause mortality comprising of 531,804 participants spanning 13.24 years, it was shown that the relative risk was proportionally reduced by 66% with at least four or more healthy lifestyle behaviours (16). In a large UK study exploring the impact of combined health behaviours on mortality, it was shown that smoking status, dietary intake, alcohol consumption and physical activity, when combined, increased risk of mortality four-fold, with demonstrable trends seen as strongest in cardiovascular causes (17).

The tendency for behaviours to cumulatively increase or decrease risk has important implications for health promotion and prevention strategies with further exploration needed to understand and define these. It is also important to examine these factors within a multiethnic population, so as to be able to ensure that any data collected is reflective of the diversity in society and that any conclusions made have validity to appropriate inform health reform, as per the DoH's Research Governance Framework for Health and Social Care (18). The current study aims to explore the clustering of lifestyle behaviours in a multi-ethnic population within Leicester City and Leicestershire County, in both primary and secondary care settings, to understand how lifestyle behaviours present, cumulate, impact upon, and associate with other behaviours and socio-demographic factors in both a healthy population and those with long-term conditions (LTCs).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over.
* Ability to read and understand English.
* Has not already completed the questionnaire.
* Able and willing to complete questionnaire.

Exclusion Criteria:

* Participant unable or unwilling to complete questionnaire.
* Under the age of 18.
* Participant has already completed the questionnaire.
* Unable to read and write in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 or over who are willing and able to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 9500 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Clustering of common lifestyle behaviours | 5 years
  To investigate the clustering of common lifestyle behaviours in a multi-ethnic population.

SECONDARY OUTCOMES:
Examine associations socio-demographic factors and lifestyle behaviours | 5 years
  To examine associations between socio-demographic factors and lifestyle behaviours, in both a healthy population and those with LTCs, to define subgroups with elevated risk of poor health outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Leicester General Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No